CLINICAL TRIAL: NCT06933992
Title: Evaluation of the Safety and Efficacy of the Chocolate Balloon Catheter in Percutaneous Transluminal Angioplasty (PTA) for Peripheral Arterial Disease (PAD): A Prospective, Multicenter, Single-Arm Observational Trial
Brief Title: Safety and Efficacy of Chocolate Balloon Catheter in Peripheral Arterial Disease (CHOCO-PAD)
Acronym: CHOCO-PAD
Status: Enrolling by invitation | Type: Observational
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: NV-001-HZFH
Record Dates: First submitted 2025-04-10; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Chocolate Balloon Catheter; Percutaneous Transluminal Angioplasty; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chocolate PTA for PAD: This cohort comprises patients with symptomatic peripheral artery disease (Rutherford class 2-5) undergoing percutaneous transluminal angioplasty (PTA) using the Chocolate balloon catheter as part of routine care. Participants will be prospectively followed for 12 months to assess target lesion patency, revascularization rates, and clinical outcomes. Inclusion criteria: age ≥18 years, de novo/restenotic lesions (≤150 mm) in native lower limb arteries, and reference vessel diameter 4-6 mm.
  Interventions: Device: Chocolate PTA Balloon Catheter

INTERVENTIONS:
Device: Chocolate PTA Balloon Catheter — The Chocolate PTA balloon catheter is a nitinol-constrained percutaneous transluminal angioplasty balloon designed to minimize vessel trauma during treatment of peripheral arterial lesions. The device is used according to its standard indications and instructions for use in patients with symptomatic peripheral artery disease.

SUMMARY:
This study aims to learn about the long-term safety and effectiveness of the Chocolate Balloon Catheter in patients with blocked leg arteries (peripheral artery disease, or PAD). The Chocolate Balloon is a special type of balloon used during minimally invasive procedures to open narrowed arteries while potentially causing less damage to the blood vessel.

The main question it aims to answer is:

Does the Chocolate Balloon keep the treated artery open after 12 months without needing repeat procedures? Patients with PAD who are already scheduled to undergo an artery-opening procedure (angioplasty) with the Chocolate Balloon as part of their standard care will answer the question about the safety and effectiveness of the Chocolate Balloon Catheter

ELIGIBILITY:
Inclusion Criteria:

* Participant or legal guardian provides written informed consent.
* Age ≥18 and ≤80 years, regardless of gender.
* De novo target lesion located in the native superficial femoral, popliteal, or infrapopliteal artery.
* Life expectancy >1 year as assessed by the investigator.
* Candidate suitable for endovascular angiography and intervention per investigator judgment.
* Willingness to undergo Chocolate Balloon Catheter PTA.

Exclusion Criteria:

* Active systemic infection or uncontrolled coagulation disorder within 14 days prior to procedure.
* Planned major amputation of the target limb (at or above the ankle).
* Renal insufficiency (MDRD eGFR ≤30 mL/min/1.73 m²) or serum creatinine ≥2.5 mg/dL within 30 days, or dialysis dependence.
* Contraindication to antiplatelet therapy (aspirin/clopidogrel), low-molecular-weight heparin, vasodilators, or contrast agents.
* Uncontrolled systemic comorbidities (e.g., severe cardiac/pulmonary/hepatic dysfunction, advanced malignancy, uncorrected coagulopathy).
* History of cerebral hemorrhage, symptomatic stroke, myocardial infarction, or gastrointestinal bleeding within 6 months.
* Pregnancy, lactation, or planned pregnancy (men or women).
* Participation in another interventional clinical trial with unmet primary endpoint.
* Investigator-determined medical, social, or psychological contraindications.
* Life expectancy <1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from patients diagnosed with symptomatic peripheral artery disease (Rutherford class 2-5) who are undergoing percutaneous transluminal angioplasty (PTA) with the Chocolate balloon catheter as part of standard care. The ages of participants range from 18 to 80 years.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Target lesion patency rate at 12 months post-procedure | From enrollment to the end of treatment at 12 months
  It is defined as the absence of restenosis (based on duplex Doppler ultrasound criteria: diameter stenosis >50% and peak systolic velocity ratio <2.5) and freedom from target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Rate of Acute Angiographic Success Defined as Core Lab-Assessed Residual Stenosis ≤30% Without Flow-Limiting Dissection (Grade D or Higher) | From enrollment to the end of treatment at 12 months
  Proportion of participants achieving successful revascularization, defined by two co-primary angiographic criteria: 1) Core laboratory-adjudicated residual stenosis ≤30%, and 2) Absence of flow-limiting dissection (Grade D or higher per NHLBI classification), assessed immediately after device deployment.
Rate of bailout stenting | From enrollment to the end of treatment at 12 months
  The proportion of cases requiring emergency stent placement due to suboptimal Chocolate balloon angioplasty results (e.g., severe dissection, recoil, or residual stenosis).
Number of Participants with Improvement in Rutherford Clinical Category from Baseline | From enrollment to the end of treatment at 12 months
  Proportion of participants achieving ≥1 category reduction in Rutherford Clinical Classification (Scale Range: 0 [asymptomatic] to 6 [major tissue loss]) at 12 months post-procedure, as assessed by blinded core lab
Freedom from clinically driven Target Lesion Revascularization (TLR) at 1, 6, and 12 months | From enrollment to the end of treatment at 12 months
  The rate of freedom from repeat revascularization (surgical or endovascular) of the target lesion due to symptoms or worsening blood flow at 1, 6, and 12 months.
Change in Ankle-Brachial Index (ABI) from Baseline | From enrollment to the end of treatment at 12 months
  Mean difference in ABI (normal range: 0.9-1.3) measurements between pre-procedure baseline and 12-month follow-up, assessed by standardized vascular laboratory protocols. Higher values indicate better perfusion.
Change in Toe-Brachial Index (TBI) from Baseline | From enrollment to the end of treatment at 12 months
  Mean difference in TBI (normal >0.6) measurements between pre-procedure baseline and 12-month follow-up, assessed by standardized vascular laboratory protocols. Higher values indicate better perfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Xiaohu, MS, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No
Due to privacy and confidentiality concerns, individual participant data (IPD) will not be shared. The data contains sensitive health information that is protected by regulations, and sharing it may compromise participant confidentiality.

REFERENCES:
- [Result] Babaev A, Zavlunova S, Attubato MJ, Martinsen BJ, Mintz GS, Maehara A. Orbital Atherectomy Plaque Modification Assessment of the Femoropopliteal Artery Via Intravascular Ultrasound (TRUTH Study). Vasc Endovascular Surg. 2015 Oct;49(7):188-94. doi: 10.1177/1538574415607361. Epub 2015 Oct 20. PMID 26490645
- [Result] Lee MS, Canan T, Rha SW, Mustapha J, Adams GL. Pooled analysis of the CONFIRM registries: impact of gender on procedure and angiographic outcomes in patients undergoing orbital atherectomy for peripheral artery disease. J Endovasc Ther. 2015 Feb;22(1):57-62. doi: 10.1177/1526602814564367. PMID 25775681
- [Result] Mintz GS, Popma JJ, Pichard AD, Kent KM, Satler LF, Chuang YC, Ditrano CJ, Leon MB. Patterns of calcification in coronary artery disease. A statistical analysis of intravascular ultrasound and coronary angiography in 1155 lesions. Circulation. 1995 Apr 1;91(7):1959-65. doi: 10.1161/01.cir.91.7.1959. PMID 7895353
- [Result] Kawaguchi R, Tsurugaya H, Hoshizaki H, Toyama T, Oshima S, Taniguchi K. Impact of lesion calcification on clinical and angiographic outcome after sirolimus-eluting stent implantation in real-world patients. Cardiovasc Revasc Med. 2008 Jan-Mar;9(1):2-8. doi: 10.1016/j.carrev.2007.07.004. PMID 18206630
- [Result] Kashyap VS, Pavkov ML, Bishop PD, Nassoiy SP, Eagleton MJ, Clair DG, Ouriel K. Angiography underestimates peripheral atherosclerosis: lumenography revisited. J Endovasc Ther. 2008 Feb;15(1):117-25. doi: 10.1583/07-2249R.1. PMID 18254670
- [Result] Allison MA, Criqui MH, Wright CM. Patterns and risk factors for systemic calcified atherosclerosis. Arterioscler Thromb Vasc Biol. 2004 Feb;24(2):331-6. doi: 10.1161/01.ATV.0000110786.02097.0c. Epub 2003 Dec 4. PMID 14656730
- [Result] Rocha-Singh KJ, Zeller T, Jaff MR. Peripheral arterial calcification: prevalence, mechanism, detection, and clinical implications. Catheter Cardiovasc Interv. 2014 May 1;83(6):E212-20. doi: 10.1002/ccd.25387. Epub 2014 Feb 10. PMID 24402839
- [Result] Fitzgerald PJ, Ports TA, Yock PG. Contribution of localized calcium deposits to dissection after angioplasty. An observational study using intravascular ultrasound. Circulation. 1992 Jul;86(1):64-70. doi: 10.1161/01.cir.86.1.64. PMID 1617791
- [Result] Hoffmann R, Mintz GS, Popma JJ, Satler LF, Kent KM, Pichard AD, Leon MB. Treatment of calcified coronary lesions with Palmaz-Schatz stents. An intravascular ultrasound study. Eur Heart J. 1998 Aug;19(8):1224-31. doi: 10.1053/euhj.1998.1028. PMID 9740344
- [Result] Laird JR, Katzen BT, Scheinert D, Lammer J, Carpenter J, Buchbinder M, Dave R, Ansel G, Lansky A, Cristea E, Collins TJ, Goldstein J, Jaff MR; RESILIENT Investigators. Nitinol stent implantation versus balloon angioplasty for lesions in the superficial femoral artery and proximal popliteal artery: twelve-month results from the RESILIENT randomized trial. Circ Cardiovasc Interv. 2010 Jun 1;3(3):267-76. doi: 10.1161/CIRCINTERVENTIONS.109.903468. Epub 2010 May 18. PMID 20484101
- [Result] Dick P, Wallner H, Sabeti S, Loewe C, Mlekusch W, Lammer J, Koppensteiner R, Minar E, Schillinger M. Balloon angioplasty versus stenting with nitinol stents in intermediate length superficial femoral artery lesions. Catheter Cardiovasc Interv. 2009 Dec 1;74(7):1090-5. doi: 10.1002/ccd.22128. PMID 19859954
- [Result] Schillinger M, Sabeti S, Loewe C, Dick P, Amighi J, Mlekusch W, Schlager O, Cejna M, Lammer J, Minar E. Balloon angioplasty versus implantation of nitinol stents in the superficial femoral artery. N Engl J Med. 2006 May 4;354(18):1879-88. doi: 10.1056/NEJMoa051303. PMID 16672699
- [Result] Yokoi Y. How should recent endovascular trials for femoropopliteal artery disease be interpreted? Cardiovasc Interv Ther. 2017 Apr;32(2):106-113. doi: 10.1007/s12928-017-0463-z. Epub 2017 Mar 1. PMID 28251562
- [Result] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Result] Rooke TW, Hirsch AT, Misra S, Sidawy AN, Beckman JA, Findeiss LK, Golzarian J, Gornik HL, Halperin JL, Jaff MR, Moneta GL, Olin JW, Stanley JC, White CJ, White JV, Zierler RE; Society for Cardiovascular Angiography and Interventions; Society of Interventional Radiology; Society for Vascular Medicine; Society for Vascular Surgery. 2011 ACCF/AHA Focused Update of the Guideline for the Management of Patients With Peripheral Artery Disease (updating the 2005 guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2011 Nov 1;58(19):2020-45. doi: 10.1016/j.jacc.2011.08.023. Epub 2011 Oct 6. No abstract available. PMID 21963765
- [Result] European Stroke Organisation; Tendera M, Aboyans V, Bartelink ML, Baumgartner I, Clement D, Collet JP, Cremonesi A, De Carlo M, Erbel R, Fowkes FG, Heras M, Kownator S, Minar E, Ostergren J, Poldermans D, Riambau V, Roffi M, Rother J, Sievert H, van Sambeek M, Zeller T; ESC Committee for Practice Guidelines. ESC Guidelines on the diagnosis and treatment of peripheral artery diseases: Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteries: the Task Force on the Diagnosis and Treatment of Peripheral Artery Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2011 Nov;32(22):2851-906. doi: 10.1093/eurheartj/ehr211. Epub 2011 Aug 26. No abstract available. PMID 21873417
- [Result] Lawall H, Huppert P, Espinola-Klein C, Zemmrich CS, Ruemenapf G. German guideline on the diagnosis and treatment of peripheral artery disease - a comprehensive update 2016. Vasa. 2017 Mar;46(2):79-86. doi: 10.1024/0301-1526/a000603. Epub 2017 Jan 27. PMID 28128018
- [Result] Zeller T. Current state of endovascular treatment of femoro-popliteal artery disease. Vasc Med. 2007 Aug;12(3):223-34. doi: 10.1177/1358863X07079823. PMID 17848483
- [Result] McDaniel MD, Cronenwett JL. Basic data related to the natural history of intermittent claudication. Ann Vasc Surg. 1989 Jul;3(3):273-7. doi: 10.1016/S0890-5096(07)60040-5. No abstract available. PMID 2673321
- [Result] Dormandy J, Mahir M, Ascady G, Balsano F, De Leeuw P, Blombery P, Bousser MG, Clement D, Coffman J, Deutshinoff A, et al. Fate of the patient with chronic leg ischaemia. A review article. J Cardiovasc Surg (Torino). 1989 Jan-Feb;30(1):50-7. PMID 2647761
- [Result] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Result] Sampson UK, Fowkes FG, McDermott MM, Criqui MH, Aboyans V, Norman PE, Forouzanfar MH, Naghavi M, Song Y, Harrell FE Jr, Denenberg JO, Mensah GA, Ezzati M, Murray C. Global and regional burden of death and disability from peripheral artery disease: 21 world regions, 1990 to 2010. Glob Heart. 2014 Mar;9(1):145-158.e21. doi: 10.1016/j.gheart.2013.12.008. PMID 25432124
- [Result] Diehm C, Schuster A, Allenberg JR, Darius H, Haberl R, Lange S, Pittrow D, von Stritzky B, Tepohl G, Trampisch HJ. High prevalence of peripheral arterial disease and co-morbidity in 6880 primary care patients: cross-sectional study. Atherosclerosis. 2004 Jan;172(1):95-105. doi: 10.1016/s0021-9150(03)00204-1. PMID 14709362
- [Result] Newman AB, Shemanski L, Manolio TA, Cushman M, Mittelmark M, Polak JF, Powe NR, Siscovick D. Ankle-arm index as a predictor of cardiovascular disease and mortality in the Cardiovascular Health Study. The Cardiovascular Health Study Group. Arterioscler Thromb Vasc Biol. 1999 Mar;19(3):538-45. doi: 10.1161/01.atv.19.3.538. PMID 10073955
- [Derived] Ye ZQ, Liu H, Fang X, Meng XH. Safety and effectiveness of the Chocolate balloon catheter in the treatment of peripheral artery disease with percutaneous transluminal angioplasty: a multicentre, prospective, observational study protocol. BMJ Open. 2025 Oct 13;15(10):e103906. doi: 10.1136/bmjopen-2025-103906. PMID 41083315
- See also: Description the protocol of the study — https://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Study Protocol — http://www.chinadrugtrials.org.cn/clinicaltrials.searchlistdetail.dhtml